CLINICAL TRIAL: NCT00261391
Title: Phase I Dose Escalation Study to Evaluate the Safety and Preliminary Efficacy of Marimastat in Patients With Disabling Malformations and No Other Treatment Options
Brief Title: Phase I Drug Trial for S/E of Marimastat in Disabling Malformations When no Other Options.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-04-052R
Record Dates: First submitted 2005-12-02; First posted 2005-12-05 (Estimated); Last update posted 2008-01-09 (Estimated); Status verified 2005-05

CONDITIONS: Vascular Anomalies
Keywords: Arteriovenous Malformation; Lymphatic Malformation; Gorham
MeSH Terms: conditions — Vascular Malformations; Arteriovenous Malformations; Lymphatic Abnormalities | interventions — marimastat

INTERVENTIONS:
Drug: Marimastat

SUMMARY:
3 patients were enrolled in each of 3 study cohorts. There three cohorts were given differing, incrementally larger doses of this phase I drug. The same safety measures are being obtained on all patients. Efficacy measures were individualized as enrolllees do not have the same underlying vascular anomaly. The study is structured to include a 24 month drug-phase and a 24 month follow-up phase. The study is now closed to enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Patient with vascular malformation causing risk of one or more of the following based on unanimous assessment of designated physicians in the multidisciplinary Vascular Anomalies Team.

  * airway/respiratory/visual/auditory/neurologic compromise;
  * high output cardiac failure;
  * life-threatening or disabling hemorrhage(cutaneous/GI/intracranial/ parenchymal/cavitary);
  * skeletal distortion/destruction/erosion;
  * life-threatening or disabling soft tissue distortion or destruction
* Patient must be felt to have failed, be unable to significantly benefit from, or be at risk for other available therapies, including surgeries, embolization, and sclerotherapy based on unanimous assessment of designated physicians in the multidisciplinary Vascular Anomalies Team.
* Patient must be felt to have one or more physical, imaging, photographic, physiologic or other measurable features that can be measured on a regular basis for preliminary evaluation of efficacy. The feature(s) must be agreed on by the designated physicians in the multidisciplinary Vascular Anomalies Team).
* Signed Patient informed consent.

Exclusion Criteria:

* Pregnancy
* Patient nursing child.
* Female patient of childbearing potential unwilling to receive contraceptive counseling and use reliable contraceptive method.
* Patient enrolled in any other clinical trial involving an investigational agent (unless approved by the designated physicians on the multidisciplinary team)
* Parent or guardian or child unwilling to provide consent or assent.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9
Dates: Start 2000-10; Study Completion 2007-10

PRIMARY OUTCOMES:
History
Physical Examination
Laboratory studies
Vital Signs
EKG
Urine studies

SECONDARY OUTCOMES:
Individualized. Change in the predetermined measure of the vascular anomaly.

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Fishman, M.D., Principal Investigator — Boston Children's Hospital
Locations (1):
- Childrens Hospital, Boston, Massachusetts, United States